CLINICAL TRIAL: NCT05323292
Title: Vitamin A Status in Patients With Vocal Fold Leukoplakia
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-1045; R01DC019357 (NIH); A539770 (Other: UW Madison); 07/01/2021 (Other: UW Madison); SMPH/SURGERY/SURGERY*OT (Other: UW Madison); 2021-1045 (Other: UW Madison)
Record Dates: First submitted 2022-03-15; First posted 2022-04-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Vitamin A; Vitamin A Deficiency; Leukoplakia; Vocal Cord Neoplasm
MeSH Terms: conditions — Vitamin A Deficiency; Leukoplakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Leukoplakia due to hyperkeratosis with dysplasia: Biopsy-confirmed diagnosis of hyperkeratosis with dysplasia.
- Leukoplakia due to hyperkeratosis with no dysplasia: Biopsy-confirmed diagnosis of hyperkeratosis with no dysplasia.
- Control group: Laryngoscopy showing no evidence of vocal fold epithelial disease.

SUMMARY:
This study will determine systemic vitamin A status and lesion histopathology of participants with vocal fold hyperkeratosis resulting in clinical leukoplakia.

DETAILED DESCRIPTION:
The investigator's overarching goal is to determine if there is a pathophysiologic rationale for vitamin A supplementation in the treatment of vocal fold hyperkeratosis. Vocal fold hyperkeratosis is an accumulation of epithelial surface keratin resulting in clinical leukoplakia. It is primarily managed using destructive techniques that risk iatrogenic injury, fibrosis, and voice impairment. Given the potential morbidity of biopsy and lesion removal, there is a need for new approaches to the prevention and treatment of vocal fold leukoplakic disorders that are non-destructive. Vitamin A is a key regulator of epithelial health and systemic vitamin A deficiency could directly contribute to hyperkeratosis. Based on vitamin A's importance to vocal fold stellate and epithelial cell biology and its direct relevance to vocal fold hyperkeratosis, this study will assess vitamin A status in participants with vocal fold hyperkeratosis. An association would suggest further study on the effects of vitamin A optimization and/or supplementation in patients with leukoplakia, as well as an adjuvant therapy in participants for whom surgical treatment is indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Ability to take oral medication.
4. At least 18 years of age.
5. Leukoplakia study groups:

   1. Leukoplakia due to hyperkeratosis with dysplasia: biopsy-confirmed diagnosis of hyperkeratosis with dysplasia.
   2. Leukoplakia due to hyperkeratosis with no dysplasia: biopsy-confirmed diagnosis of hyperkeratosis with no dysplasia.
6. Control group: Laryngoscopy showing no evidence of vocal fold epithelial disease.

Exclusion Criteria:

1. History of malignant vocal fold epithelial pathology.
2. History of metabolic or liver disorder.
3. History of anorexia or bulimia.
4. Pregnant, lactating, or planning on becoming pregnant during the study period.
5. History of >4.5 kg weight loss in the past 90 days.
6. Medical or other inability to complete an 8 hour fast.
7. Acute respiratory or gastrointestinal illness.
8. Currently incarcerated.
9. Impaired decision-making capacity.
10. No or limited English speaking ability; illiterate or low-literacy ability.
11. Profound visual or hearing impairment that limits written or verbal communication.
12. Status relationship with a member of the study team.
13. Not suitable for study participation due to other reasons at the discretion of the investigators.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified from the active caseloads of speech-language pathologists or otolaryngologists. During a routine clinical encounter, a member of the clinical team will inform potential participants of the research opportunity.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin A liver reserves | 14 days
  Total vitamin A liver concentration determined using retinol stable isotope dilution (μmol/g)

SECONDARY OUTCOMES:
Serum retinol | Baseline
  Serum retinol concentration (μmol/L)
Serum retinyl esters | Baseline
  Serum retinyl esters concentration (μmol/L)
Serum carotenoids | Baseline
  Serum carotenoid concentrations (μmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Welham, PhD, CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No